CLINICAL TRIAL: NCT00208026
Title: Exploratory Safety and Systemic Absorption of Elidel (Pimecrolimus) 1% Cream for the Treatment of Netherton Syndrome
Brief Title: Safety Study of Elidel (Pimecrolimus) 1% Cream to Treat Netherton Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Albert Yan, Principal Investigator, Children's Hospital of Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-11-4063
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Netherton Syndrome
MeSH Terms: conditions — Netherton Syndrome | interventions — pimecrolimus; WAS protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pimecrolimus 1% Cream (Experimental): Treatment with drug/Elidel. Single arm-open-label treatment arm. A Pilot Study of the Efficacy and Safety of Pimecrolimus Cream 1% for the Treatment of Netherton Syndrome:
  Interventions: Drug: Pimecrolimus 1% Cream

INTERVENTIONS:
Drug: Pimecrolimus 1% Cream — Open label single arm
  Other Names: Elidel; Eczema

SUMMARY:
Netherton syndrome is a genetic condition that can result in abnormal skin functioning. People with this condition often have red and scaling skin; sparse or short hair; and problems with absorption of medicines or chemicals that are applied to the skin. If these chemicals are absorbed at a high level, they may cause health problems. Elidel (pimecrolimus) is a new medicine that is available as a cream. It has been shown to help improve the appearance of the skin in patients with another skin condition known as atopic dermatitis, and is approved by the United States (US) Food and Drug Administration for use in children with mild to moderate atopic dermatitis. The purpose of this study is to determine if Elidel is safe, to see whether the medication is absorbed through the skin, and to see if side effects are associated with its use in children with Netherton syndrome.

DETAILED DESCRIPTION:
Patients with Netherton syndrome, a rare genodermatosis, manifest a chronic, eczematous dermatitis with erythema and scaling that is often recalcitrant to conventional therapy with emollients and topical corticosteroids. These patients display an altered epidermal barrier with increased permeability to topical agents and are therefore susceptible to evaporative transepidermal water loss and infection. Topical therapy with the calcineurin inhibitors tacrolimus and pimecrolimus has been demonstrated to improve the skin integrity and the quality of life of patients with several chronic dermatoses, including atopic dermatitis. As a result of the underlying skin barrier dysfunction, however, the possibility of significant systemic absorption and resultant side effects is a concern when these agents are used in patients with Netherton syndrome. Experience with topical tacrolimus 0.1% ointment for patients with Netherton syndrome has demonstrated both marked efficacy as well as significant systemic absorption of the drug in this patient population. Use of topical pimecrolimus in patients with Netherton syndrome has not been reported to date. Investigation of the extent of systemic absorption and side effects will help to define the safety and efficacy profile of topical pimecrolimus in patients with Netherton syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Netherton syndrome
* Normal laboratory values within 3 months prior to enrollment
* Signed written informed consent
* Willingness and ability to comply with the study requirements
* For women of childbearing age, negative urine pregnancy test at enrollment and then monthly thereafter; women of childbearing age who are not abstinent must use contraception.

Exclusion Criteria:

* Clinically significant physical examination or laboratory abnormalities
* Clinical evidence of liver disease or liver injury as documented by abnormal liver function tests
* Symptoms of a significant acute illness in the 30 week period preceding the start of treatment
* Patients with known serious adverse reactions or hypersensitivity to macrolides or calcineurin inhibitors or with known hypersensitivity to any of the ingredients of the study medication or history of adverse reactions to the anesthetic product used for blood draws
* Topical tacrolimus or Elidel within 2 weeks prior to dosing
* Systemic steroid, systemic tacrolimus, or any immunosuppressant within 1 month prior to dosing
* Phototherapy within 1 month prior to dosing
* Use of inhibitors of Cytochrome P450 3A4 (CYP3A4) iso-enzyme within 2 weeks prior to dosing
* Topical steroids or other topical therapy (except tacrolimus) may be used up to the day of 1st application of Elidel; however, treatment must be discontinued during the treatment period. Topical treatment of corticosteroids may resume immediately after the treatment period or in case an alert value has been exceeded and the Elidel treatment will be continued only on the face and neck.
* Participation in any clinical trials within 2 months prior to dosing
* History or clinical evidence of cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematologic, neurologic disease, or any disease other than Netherton syndrome, that may put the subject at undue risk. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs.
* History of presence of malignancy or lymphoproliferative disease
* Presence of any viral or fungal or untreated bacterial skin infection
* Known HIV positivity or active hepatitis B or C
* History of immunocompromise
* No vaccines containing live viruses are to be administered during the study period.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2005-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert C Yan, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Yan AC, Honig PJ, Ming ME, Weber J, Shah KN. The safety and efficacy of pimecrolimus, 1%, cream for the treatment of Netherton syndrome: results from an exploratory study. Arch Dermatol. 2010 Jan;146(1):57-62. doi: 10.1001/archdermatol.2009.326. PMID 20083693
- See also: Children's Hospital of Philadelphia — http://www.chop.edu
- See also: Foundation for Ichthyosis and Related Skin Types — http://www.scalyskin.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label,single-arm study to investigate the safety profile of topical pimecrolimus cream.
  Patients meeting the criteria for diagnosis of Netherton Syndrome were enrolled over a period of 3 years, from September 2005 through March 2008. The study was conducted in my medical office within The Children's Hospital of Philadelphia.
Pre-assignment Details: The eligibility was for male and female patients aged 2 to 18 years.They were required to have normal laboratory values within 3 months prior to enrollment. A 4 week washout period was required for systemic steroid, tacrolimus, immunosuppressives, phototherapy, and inhibitors of Cytochrome. 2 week washout for Isoenzyme,tacrolimus and pimecrolimus.
Groups:
- Elidel (Pimecrolimus) 1% Cream: Treatment with drug/Elidel.Single arm-open-label treatment arm. A Pilot Study of the Efficacy and Safety of Pimecrolimus Cream 1% for the Treatment of Netherton Syndrome:
Period: Overall Study
Arm/Group | Elidel (Pimecrolimus) 1% Cream
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Elidel (Pimecrolimus) 1% Cream
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Blood Pimecrolimus Levels
Description: At each scheduled visit, blood concentration of pimecrolimus were obtained. This value reflects the amount of pimecrolimus in the blood. This is measured directly from the blood and provides an estimate of the degree of absorption of the treatment medication through the skin into the blood.
Time Frame: Each visit up to 18 months: Study Days 1, 7, 14, 28, 56, 84, 175, 360, and 520
Measure: Number; unit: ng/mL
Groups:
- Patient 1; Patient 2; Patient 3: Treatment with drug/Elidel. Single arm-open-label treatment arm. A Pilot Study of the Efficacy and Safety of Pimecrolimus Cream 1% for the Treatment of Netherton Syndrome:
  Pimecrolimus 1% Cream: Open label single arm
Arm/Group | Patient 1 | Patient 2 | Patient 3
Number analyzed (Participants) | 1 | 1 | 1
ng/mL
  Day 1 | 0 | 0 | 0.312
  Day 7 | 1.260 | 0.625 | 3.630
  Day 14 | 0.821 | 0.421 | 3.930
  Day 28 | 0.592 | 0.311 | 7.080
  Day 56 | 0.743 | 0.182 | 3.920
  Day 84 | 0.390 | 0.368 | 5.010
  Day 175 | 0.470 | 0.484 | 2.060
  Day 360 | 0.388 | 0.247 | 4.280
  Day 520 | 0.224 | 0.170 | 6.140

ADVERSE EVENTS:
Time Frame: During the 18 month study, all 3 patients were evaluated throughout the study.
Description: No serious adverse events were reported.
Arm/Group | Elidel (Pimecrolimus) 1% Cream
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
There were no early termination for any of the subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No